CLINICAL TRIAL: NCT00511329
Title: Growth and the Effect of Genotropin in Chronically Ill Children With Juvenile Rheumatoid Arthritis and With Crohn's Disease
Brief Title: Growth Hormone in Children With Juvenile Rheumatoid Arthritis (JRA) and With Crohn's Disease
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: PI left the institution
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GA628132
Record Dates: First submitted 2007-08-02; First posted 2007-08-03 (Estimated); Results first posted 2018-04-12 (Actual); Last update posted 2018-04-12 (Actual); Status verified 2018-03

CONDITIONS: Arthritis, Juvenile Rheumatoid; Crohn Disease
Keywords: growth hormone; short stature; growth failure; chronic illness
MeSH Terms: conditions — Arthritis, Juvenile; Crohn Disease; Dwarfism; Failure to Thrive; Chronic Disease | interventions — Human Growth Hormone; WW Domain-Containing Oxidoreductase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Somatropin (Experimental)
  Interventions: Drug: somatropin [rDNA origin] for injection

INTERVENTIONS:
Drug: somatropin [rDNA origin] for injection — Genotropin will be started at 0.3 mg/kg/week administered by daily subcutaneous injection. Doses will be increased by weight at each visit. Additionally, we will monitor IGF-1 levels at month 3, and 6 and adjust the Genotropin dose to maintain IGF-1 levels in the 50th -75th percentile for ages.
  Other Names: Genotropin

SUMMARY:
The investigators hypothesize that the anabolic effects of Genotropin (somatropin) will improve the height and weight of children with inflammatory based chronic illness who have failed to grow despite receiving adequate nutrition. The investigators will test the hypothesis by treating 32 chronically ill children (16 JRA and 16 Crohn's) with growth hormone (GH) for 12 months and comparing them to baseline.

DETAILED DESCRIPTION:
1. To determine the effect of GenotropinTM on height, height velocity, body weight and lean body mass. Growth records from previous years will be assessed to determine growth velocity and weight gain. We will measure height and weight during the study using a standardized stadiometer and scale. These parameters will be converted to Z scores (GenenCalcTM, Genentech). Lean body mass (LBM) will be measured by DXA every six months. This specific aim tests the hypothesis that GH significantly improves height, height velocity, weight, weight velocity and LBM in chronically ill children who have grown poorly despite adequate nutritional rehabilitation.
2. To determine the effect of GenotropinTM on whole body protein turnover (WBPT), IGF-1 levels and cytokines. Utilizing the stable isotope 1-[13C] leucine, we will measure WBPT. Measurements of WBPT will be correlated with LBM and changes in height and weight velocity. This data will be compared to that from age matched normal children (archival data maintained by the PI). We will measure IGF-1 and the cytokines TNF-α, IL-6 and IL-10 at baseline and very six months. These measures will be correlated with height and weight velocity and IGF-1 levels. Cytokine levels will also be correlated with protein catabolism. This specific aim tests the hypothesis that chronically ill children have increased catabolism, caused by high levels of circulating cytokines and low levels of IGF-1, and that these abnormalities improve with GenotropinTM.
3. Evaluation of bone mineral content (BMC) and bone turnover. At baseline and every six months we will measure BMC of the whole body, hip and spine using DXA. Results will be compared to those from age-matched normal children whose results are archived in the body composition laboratory of Dr. Ken Ellis (Children's Nutrition Research Center, Houston). At baseline and every six months we will also measure bone mineral turnover markers including: osteocalcin, bone specific alkaline phosphatase activity, and deoxypyridinoline. All findings will be related to cytokine levels and to use of glucocorticoids. This specific aim tests the hypothesis that bone density is low in chronically ill children secondary to increased osteoclast activity correlating with elevated cytokine levels.

ELIGIBILITY:
Inclusion Criteria:

1. Referral for continued poor growth (growth velocity less than the 25th percentile)
2. Height less than the 10th percentile
3. Weight less than the 10th percentile compared to age and gender- matched normal values.

Exclusion Criteria:

1. Previous diagnosis with diabetes, chronic fevers (temp > 101.5) or chronic bacterial infection
2. Previous treatment with GH
3. Bone age > 17

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2007-08; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dana S Hardin, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Columbus Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Background] Bechtold S, Ripperger P, Muhlbayer D, Truckenbrodt H, Hafner R, Butenandt O, Schwarz HP. GH therapy in juvenile chronic arthritis: results of a two-year controlled study on growth and bone. J Clin Endocrinol Metab. 2001 Dec;86(12):5737-44. doi: 10.1210/jcem.86.12.8083. PMID 11739431
- [Background] Mauras N, George D, Evans J, Milov D, Abrams S, Rini A, Welch S, Haymond MW. Growth hormone has anabolic effects in glucocorticosteroid-dependent children with inflammatory bowel disease: a pilot study. Metabolism. 2002 Jan;51(1):127-35. doi: 10.1053/meta.2002.28972. PMID 11782884
- [Background] Hardin DS, Ellis KJ, Dyson M, Rice J, McConnell R, Seilheimer DK. Growth hormone decreases protein catabolism in children with cystic fibrosis. J Clin Endocrinol Metab. 2001 Sep;86(9):4424-8. doi: 10.1210/jcem.86.9.7822. PMID 11549686
- [Background] Hardin DS, Rice J, Doyle ME, Pavia A. Growth hormone improves protein catabolism and growth in prepubertal children with HIV infection. Clin Endocrinol (Oxf). 2005 Sep;63(3):259-62. doi: 10.1111/j.1365-2265.2005.02331.x. PMID 16117811
- [Background] Hardin DS, Adams-Huet B, Brown D, Chatfield B, Dyson M, Ferkol T, Howenstine M, Prestidge C, Royce F, Rice J, Seilheimer DK, Steelman J, Shepherds R. Growth hormone treatment improves growth and clinical status in prepubertal children with cystic fibrosis: results of a multicenter randomized controlled trial. J Clin Endocrinol Metab. 2006 Dec;91(12):4925-9. doi: 10.1210/jc.2006-1101. Epub 2006 Oct 3. PMID 17018651

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: PI left institution suddenly in 2010 and studies were closed. Study records for participants cannot be located and possibly have been destroyed.
Period: Overall Study
Arm/Group | Somatropin
Started | 0
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: PI left institution suddenly in 2010 and studies were closed. Study records for participants cannot be located and possibly have been destroyed.
Arm/Group | Somatropin
Number analyzed (Participants) | 0
Age, Categorical
Age, Continuous [unit: years]
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome Variables Will be Height and Weight Z Score.
Time Frame: 12 months
Population: as for baseline characteristics
Arm/Group | Somatropin
Number analyzed (Participants) | 0

2. Secondary Outcome: Secondary Outcome Variables Will Include Change in Lean Body Mass, Change in Bone Mineral Content, Change in Inflammatory Mediated Cytokine Levels and Change in Bone Turnover.
Time Frame: 12 months
Population: as for baseline characteristics
Arm/Group | Somatropin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: PI left institution suddenly in 2010 and studies were closed. Study records for participants cannot be located and possibly have been destroyed.
Arm/Group | Somatropin
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes